CLINICAL TRIAL: NCT03072108
Title: Effect of Oleuropein-based Dietary Supplement (Bonolive™) Versus Placebo on Knee Joint Functionality and Cartilage Catabolism in Ageing Population
Brief Title: Dietary Supplement for Joint: the OLE Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Artialis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 15.16.CLI
Record Dates: First submitted 2017-01-31; First posted 2017-03-07 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Knee Discomfort; Knee Pain
MeSH Terms: interventions — Bonolive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bonolive (Experimental)
  Interventions: Dietary Supplement: Bonolive
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bonolive — 2 caps per day of Bonolive
  Arms: Bonolive
Dietary Supplement: Placebo — 2 caps per day of Placebo
  Arms: Placebo

SUMMARY:
This clinical study evaluates if the oral administration of Bonolive can contribute to the improvement of functionnality in healthy elderly people with knee discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 55 years of age
* BMI between 18.5 and 29.9 kg/m2 (normo and overweight)
* Moderate knee pain (the most painful knee is considered)
* Able to follow the instructions of the study
* Able to perform physical tests
* Having signed an informed consent

Exclusion Criteria:

Related to knee

* Recent trauma (< 1 month) of the knee responsible of the symptomatic knee
* Subject with knee/joint surgery/replacement and ACL (Cross Ligament) injury in the target knee
* Concurrent articular disease interfering with the evaluation of pain such as articular dysplasia, aseptic osteonecrosis, acromegaly, Paget's disease, hemophilia, hemochromatosis, chondromatosis, villonodular synovitis of the knee, seronegative spondyloarthropathy, rheumatoid arthritis, gouty arthritis , infectious arthritis, radiculalgia in the lower limbs, arteritis
* Prosthesis in the target knee
* Diagnosed arthrosis eligible to knee/joint surgery/replacement

Related to treatments

* Analgesics to manage knee pain 24h before inclusion visit
* Corticosteroids injection in the target knee in the month preceding inclusion
* Hyaluronan injection in the target knee in the last 6 months
* Oral corticotherapy ≥ 5mg/day in the last 3 months
* Symptomatic slow-acting drugs (SYSADs) treatment (Chondroitin, diacerein, glucosamine, soy and avocado unsaponifiables) in the last 3 months
* Other dietary supplements used for articular disorders in the last 3 months
* An anticipated need for the duration of the trial of corticosteroids or hyaluronan injection, oral corticotherapy, arthroscopy, analgesics other than listed as rescue treatments, which are forbidden during the trial
* Arthroscopy in the last 6 months
* Allergy or contra-indication to Oleuropein, to maltodextrin or any ingredient present in the product, or intolerance to rescue treatment (Paracetamol and NSAIDs)
* Treatments based on strontium ranelate, bisphosphonates, selective estrogen-receptor modulator (SERM) and parathormone (PTH) during the year before inclusion

Related to associated diseases

* Severe and uncontrolled diseases (liver or renal failure, lung/heart severe disease, Parkinson, progressive malignant neoplasia or in remission for less than 5 years, HIV, etc.)
* Lower or upper extremity surgery or fracture in the last 3 months
* Anticipated need for any surgical or other invasive procedure during the trial including prosthesis in the target knee
* Swallowing disorder

Related to patients

* Close collaborators to the investigational team, the study coordinator (Artialis) or to the Sponsor (Nestlé)
* Currently participating or having participated in another therapeutic clinical trial in the three previous months
* Having made a blood donation in the past month
* Under guardianship or judicial protection
* Pregnancy, breastfeeding, planned conception
* Premenopausal women or women without tubal ligation or contraception.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2016-06-24 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effect of investigational product after 6 months of supplementation | From Baseline to 6 months of product administration and compared to Placebo
  KOOS (Knee injury and Osteoarthritis Outcome Score)
Evaluation of the effect of investigational product after 6 months of supplementation | From Baseline to 6 months of product administration and compared to Placebo
  Biomarker of cartilage breakdown (Coll2.1-NO2)

SECONDARY OUTCOMES:
Evaluation of the effect of investigational product | From Baseline to 6 months of product administration and compared to Placebo
  Knee pain VAS score at rest and at walking
Evaluation of the effect of investigational product | From Baseline to 6 months of product administration and compared to Placebo
  OARSI core set of performance-based tests

OTHER OUTCOMES:
Evaluation of food habits and frequency using patient-reported questionnaire | From the date of inclusion until end of study, on a monthly basis, up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No